CLINICAL TRIAL: NCT05423054
Title: The Effect of Abdominal Massage on Gastrointestinal Outcomes Among Critically Ill Patients Receiving Enteral Feeding
Brief Title: Effect of Abdominal Massage on Gastrointestinal Outcomes Among Critically Ill Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Noura Mohamed Othman, Demonstrator in Critical Care and Emergency Nursing Department, Faculty of Nursing, Mansoura University, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P.0236
Record Dates: First submitted 2022-05-29; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Abdominal Massage

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- abdominal massage group (Experimental): * Patients will be positioned on their back while their knees will be flexed.
  * Each patient will receive a 15-minute abdominal massage intervention half an hour before enteral feeding twice per day and the interval between two massages is 2 hours for consecutive 3 days.
  * The PR will be standed on the right side of the patient during the massage practice.
  * The abdominal massage technique will be delivered to each patient in four consecutive strokes including stroking, effleurage, kneading and vibration.
  Interventions: Other: Abdominal massage
- Control group (No Intervention): The Control group will receive routine care in the intensive care unit

INTERVENTIONS:
Other: Abdominal massage — * Patients will be positioned on their back while their knees will be flexed.
  * Each patient will receive a 15-minute abdominal massage intervention half an hour before enteral feeding twice per day and the interval between two massages is 2 hours for consecutive 3 days.
  * The PR will be standed on the right side of the patient during the massage practice.
  * The abdominal massage technique will be delivered to each patient in four consecutive strokes including stroking, effleurage, kneading and vibration.
  Arms: abdominal massage group

SUMMARY:
This study aims to investigate the effect of abdominal massage on gastrointestinal outcomes among critically ill patients receiving enteral feeding.

DETAILED DESCRIPTION:
Enteral feeding has a vital role in the care of critically ill patients. It is considered a routine patients care in intensive care units. Enteral feeding is also a medical treatment as well as a part of nursing care. It is the preferred route of nutritional support in patients who are incapable of volitional intake. Additionally, it helps to stimulate peristaltic movements of the digestive system, improves blood supply, strengthens the immune system, improves recovery, and reduces physiological stress.

There are many complications associated with enteral feeding that can lead to an interruption of the feeding process, including gastrointestinal disorders, mechanical problems, fluid-electrolyte imbalance, and metabolic complications. Feeding intolerance is the most main digestive complication including nausea, vomiting, diarrhea, excess gastric residual volume, abdominal distention, and constipation.

Aspiration is also a significant side effect of delayed gastric emptying and increased GRV among CIPs. The Society of Critical Care Medicine and the American Society for Parenteral and Enteral Nutrition has recognized aspiration as one of the mutual complications of enteral feeding that should be evaluated before and during the feeding process. Consequently, prolonged ICU stays, and increased duration of mechanical ventilation, and mortality rate are side effects of feeding intolerance and aspiration. Additionally, abdominal massage is one of the complementary and alternative medicine which is significantly grown in recent years. Furthermore, it is an inexpensive, non-invasive intervention, and free from harmful side effects. Besides, it can increase the number of intestinal movements and lead to easier food movement along the gastrointestinal tract. In addition, it allows contraction of the diaphragm more fully, increases the capacity of the lung, and strengthens breathing.

ELIGIBILITY:
Inclusion Criteria:

* All patients who are Full Outline of Unresponsiveness (FOUR) score is from 0-14 admitted to the previous ICUs who have nasogastric tube and within the first 24 hours from beginning enteral feeding will be included in the study.
* Age: adult CIPs ≥ 18 years.
* Gender: males and females.
* Negative gastric pH and glucose strip.

Exclusion Criteria:

* Gastric intolerance (delayed gastric empty).
* Patients who suffered from spinal cord injury, could not be properly positioned for massage due to severe trauma.
* Patients receiving prokinetic medications (to avoid interfering with the massage effects).
* Patients who have contraindications to abdominal massage such as ascites, abdominal aortic aneurysm, ileus, diarrhea, recent abdominal surgery, bleeding of GI, abdominal tumor, and undergoing radiotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-06-20 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Investigate the effect of abdominal massage on amount of gastric residual volume among critically ill patients receiving enteral feeding | 3 days
  Change amount of gastric residual volume in milliliters
Investigate the effect of abdominal massage on abdominal circumference among critically ill patients receiving enteral feeding | 3 days
  Change abdominal circumference in Centimeter
Investigate the effect of abdominal massage on the occurrence of vomiting, constipation, and aspiration among critically ill patients receiving enteral feeding | 3 days
  Change occurrence of vomiting, constipation, and aspiration among critically ill patients receiving enteral feeding